CLINICAL TRIAL: NCT03165903
Title: Habitual and Neurocognitive Processes in Adolescent Obesity Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claremont Graduate University (Other)
Responsible Party: Principal Investigator, Kim D. Reynolds, Professor, Claremont Graduate University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U01HL097839 (NIH)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Behavioral Intervention; Obesity Prevention; Diet; Adolescents
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cue and Implementation-Intention (Experimental): Families from a school assigned to Cue and Implementation Intention-Based Intervention received an intervention targeting increased levels of healthy snacking and reduced levels of sugar sweetened beverage consumption.
  Interventions: Behavioral: Cue and Implementation Intention-Based Intervention
- Control Arm (Other): Families that were from a school assigned to Control received an intervention on sun safety that consisted of a 10-minute meeting with a trained Health Coach, 2 generic newsletters, an email, and a text message.
  Interventions: Behavioral: Control arm

INTERVENTIONS:
Behavioral: Cue and Implementation Intention-Based Intervention — Families from a school assigned to Cue and Implementation Intention-Based Intervention received an intervention targeting increased levels of healthy snacking and reduced levels of sugar sweetened beverage consumption. The intervention consisted of a 90-minute meeting with a trained Health Coach, two 20-minute phone calls, 4 tailored newsletters, and a series of emails and text messages. Cues for snacking and sweetened beverage consumption were removed or relocated and implementation-intentions were created to trigger alternative behaviors to snacking and sweetened beverage consumption in the presence of cues. Both interventions were delivered over 3-10 weeks depending on the self-directed pace of the participants. All participants completed a follow-up assessment 3 months after consent.
  Arms: Cue and Implementation-Intention
Behavioral: Control arm — Families that were from a school assigned to Control received an intervention on sun safety that consisted of a 10-minute meeting with a trained Health Coach, 2 generic newsletters, an email, and a text message. Both interventions were delivered over 3-10 weeks depending on the self-directed pace of the participants. All participants completed a follow-up assessment 3 months after consent.
  Arms: Control Arm

SUMMARY:
The study tested an intervention that used a cue-removal and implementation intentions based strategy to change habitual dietary behaviors. The intervention was evaluated using a randomized experimental design that consisted of two conditions including (1) a control condition or (2) a cue and implementation intention-based intervention. High schools (N=22) were randomly assigned to one of the two conditions. Families (N=187), with a family defined as an adolescent and one participating parent, were recruited from within the 22 schools. All of the families from each school were assigned to the same condition.

Families that were eligible for the study and that were interested in participating scheduled an appointment to complete informed consent. After written parental consent and youth assent was obtained, the participants had their height and weight measured and completed a series of questionnaires programmed on laptops. In addition, the adolescent took part in a 24 Hour Dietary Recall Assessment. The family was also informed that a second 24 Hour Dietary Recall Assessment would be administered to the adolescent over the phone in approximately 3-14 days.

Families that were from a school assigned to the control condition received an intervention on sun safety that consisted of a 10-minute meeting with a trained Health Coach, two generic newsletters, an email, and a text message. Families from a school assigned to the cue- and implementation intentions condition received an intervention on healthy snacking and the reduction of sugar sweetened beverage consumption that consisted of a 90-minute meeting with a trained Health Coach, two 20-minute phone calls, four tailored newsletters, and a series of emails and text messages. Both of these interventions were delivered over a period of 3-10 weeks depending on the self-directed pace of the participants. All participants were then asked to complete a follow-up assessment appointment three months after their original consenting appointment. Our hypotheses focused on dietary behaviors and stated that adolescents assigned to the cue-removal and implementation intentions intervention would consume significantly fewer daily servings of high fat snacks, high sugar snacks, and sugar sweetened beverages than adolescents in the control condition.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria for adolescents included being English-speaking,
* between the ages of 14 and 17,
* free of major illness,
* not receiving clinical treatment for obesity,
* possessing a cell phone with text messaging capability.

Exclusion Criteria:

* failure to meet inclusion criteria

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sugar-Sweetened Beverage servings/day | 3 months
  Change in Sugar-Sweetened Beverage consumption after intervention, through survey administration
Salty Snack servings/day | 3 months
  Change in Salty Snack consumption after intervention, through survey administration
Sweet Snacks servings/day | 3 months
  Change in Sweet Snack consumption after intervention, through survey administration

CONTACTS AND LOCATIONS:
Overall Officials: Kim D Reynolds, PhD, Principal Investigator — Claremont Graduate University

IPD SHARING:
Plan to Share IPD: Yes
The adolescent baseline and follow-up and parent's baseline and follow up data will be available. The baseline/follow up surveys and data dictionaries will be available. The data are currently available from the Principal Investigator, and the study team is working toward placement of the materials with a national data sharing center.